CLINICAL TRIAL: NCT02408783
Title: Validation of a New Simplified Score for Assessing Gestational Age of Newborns in Community
Brief Title: Simplified Gestational Age Score
Acronym: SGAS
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Massachusetts General Hospital (Other); Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Sponsor
Other Study IDs: CP SGA
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Gestational Age and Weight Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A large number of mothers are uncertain of the date of their last menstrual period and where there is a high incidence of small-for-dates babies, there is a real need for a method of estimating gestational age that is both rapid and accurate for early referral and management of preterm newborns to reduce their mortality and morbidity. The National Family Health Survey 2005-06 reports that the proportion of low birth weight babies (LBW) in India is 22%. Of these LBW babies, the proportion of prematurity is not known in the survey as it is difficult to measure gestational age of the newborn due to lack of reliable and valid scores with ease of use at the primary health centers. Different scores to assess maturity have been developed namely New Ballard score, Dubowitz score and Meharban Singh score. It is not known whether these scores have regional, geographical, racial or ethnic robustness. It has also been found that these scores tend to overestimate newborns > 37 weeks and underestimate those >32 and < 37 weeks. The investigators conducted a cross sectional study to validate three neonatal gestational age (GA) assessment scores namely New Ballard, Dubowitz and Meharban Singh with the reference standard i.e. GA assessed by LMP using Naegeles rule and validated by gestational ages also assessed by at least one ultrasound (GA-LMP), in Indian newborns delivered at a tertiary hospital. The investigators derived a new "Simplified Gestational Age Score" (SGAS) using the best applicable items from the three validated scores and assessed its accuracy with the reference standard (GA-LMP). This score has only 4 items (posture, skin texture, breast and genital assessment) and community health workers can be trained in implementing SGAS due to its simplicity. The investigators propose a study in the GN sites to validate this simplified method of assessment of the GA using our SGAS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Delivery
* Live Birth
* Correct LMP Known
* At least one USG of Ante-natal Period Reporting GA Available
* GA by LMP and USG within one week of each other
* Available for Examination up to 24 Hours of Birth
* Informed Consent Given

Exclusion Criteria:

* Menstrual Cycle Irregular
* Twin Babies
* Birth Asphyxia/ baby required Bag and Mask ventilation
* Major Congenital Anomaly
* Signs of neurological depression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Global Network Nagpur, India site will select 5 distinct Health Facilities with an average of more than 300 deliveries per year. All women who deliver in the study Health Facilities will be eligible for study enrolment after fulfilling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15920 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Validation of score tool | All gestational age assessments will be taken within 24 hours of birth
  Validity of Simplified Gestational Age Score (SGAS) when used by the ANMs and verified using the GA assessed using LMP and Sonologic GA.

SECONDARY OUTCOMES:
Variability of observer use of score tool | All gestational age assessments will be taken within 24 hours of birth
  The inter observer variability in the GA assessed by the ANM and the RO

CONTACTS AND LOCATIONS:
Overall Officials: Archana Patel, MD, Principal Investigator — Lata Medical Research Foundation
Locations (3):
- India (3):
  - Daga Memorial, Nagpur
  - GH Bhandara, Nagpur
  - GH Wardha, Nagpur

REFERENCES:
- [Background] International Institute for Population Sciences (IIPS) and ORC Macro (2006). National Family Health Survey (NFHS-3), 2005-06: India. Mumbai: IIPS.
- [Background] Barbara JS, Ira AC. The high risk infant. Cha. 97.2 Premature and intrauterine growth retardation. Nelson's Textbook of Pediatrics 18th ed. 1:701-2.
- [Background] Ballard JL, Khoury JC, Wedig K, Wang L, Eilers-Walsman BL, Lipp R. New Ballard Score, expanded to include extremely premature infants. J Pediatr. 1991 Sep;119(3):417-23. doi: 10.1016/s0022-3476(05)82056-6. PMID 1880657
- [Background] Dubowitz LM, Dubowitz V, Goldberg C. Clinical assessment of gestational age in the newborn infant. J Pediatr. 1970 Jul;77(1):1-10. doi: 10.1016/s0022-3476(70)80038-5. No abstract available. PMID 5430794
- [Background] Singh M, Razdan K, Ghai OP. Modified scoring system for clinical assessment of gestational age in the newborn. Indian Pediatr. 1975 Apr;12(4):311-6. No abstract available. PMID 1158500
- [Background] Williams obstetrics. Ed. 22nd Ch. 8. Naegele rule Page 208.
- [Derived] Patel AB, Kulkarni H, Kurhe K, Prakash A, Bhargav S, Parepalli S, Fogleman EV, Moore JL, Wallace DD, Hibberd PL. Early identification of preterm neonates at birth with a Tablet App for the Simplified Gestational Age Score (T-SGAS) when ultrasound gestational age dating is unavailable: A validation study. PLoS One. 2020 Aug 31;15(8):e0238315. doi: 10.1371/journal.pone.0238315. eCollection 2020. PMID 32866202
- [Derived] Patel AB, Kurhe K, Prakash A, Bhargav S, Parepalli S, Fogleman EV, Moore JL, Wallace DD, Kulkarni H, Hibberd PL. Early Identification of Preterm Neonates at Birth With a Tablet App for the Simplified Gestational Age Score (T-SGAS) When Ultrasound Gestational Age Dating Is Unavailable: Protocol for a Validation Study. JMIR Res Protoc. 2019 Mar 12;8(3):e11913. doi: 10.2196/11913. PMID 30860484